CLINICAL TRIAL: NCT00806624
Title: A Phase 2, Randomized, Parallel Group, Multi-Center, Multi-National Study for the Evaluation of Safety and Efficacy of Two Fixed Dosages of DU-176b in Subjects With Non-Valvular Atrial Fibrillation
Brief Title: DU-176b Phase 2 Dose Finding Study in Subjects With Non-valvular Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DU176b-C-J226
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2015-01

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — edoxaban; Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 (Experimental): DU-176b tablets: high-dose
  Interventions: Drug: DU-176b tablets
- 3 (Active Comparator): Warfarin tablets
  Interventions: Drug: Warfarin tablets
- 1 (Experimental): DU-176b tablets: low-dose
  Interventions: Drug: DU-176b tablets

INTERVENTIONS:
Drug: DU-176b tablets — DU-176b tablets taken once daily for up to 3 months
  Arms: 1
Drug: DU-176b tablets — DU-176b tablets taken once daily for up to 3 months
  Arms: 2
Drug: Warfarin tablets — Warfarin tablets taken once daily for up to 3 months
  Arms: 3

SUMMARY:
This study will be conducted in male and female subjects aged 18 to 80 years, inclusive, with non-valvular AF and a CHADS2 Score of at least 1. Subjects will be treated on an outpatient basis. The subjects will be allocated randomly to the open-label warfarin or any double-blind DU-176b dosages. DU-176b will be administered orally for 12 weeks at two fixed doses. Warfarin will be used as active control. Warfarin dosing will be managed and monitored by the Investigator with the dose adjusted to achieve an INR of 2.0 to 3.0, inclusive. The primary endpoints are incidence of major, clinically relevant non-major and minor bleeding events (all bleeding).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 to 80 years of age
* Non-valvular AF supported by abnormal ECG documented for two times (interval of more than 1 week) within 6 months prior to randomization.
* CHADS2 Score of at least 1.

Exclusion Criteria:

* Subjects with mitral valve disease
* Subjects with previous valvular heart surgery
* Contraindication for anticoagulants
* Conditions associated with high risk of bleeding
* Acute coronary syndromes (ACS), percutaneous coronary intervention (PCI), MI, stroke, transient ischemic attack (TIA) or coronary artery/cardiac/other major surgery within the previous 30 days
* Active infective endocarditis or life-expectancy < 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Hong Kong, China
- Singapore, Singapore
- Seoul, South Korea
- Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Groups:
- DU176b 30mg: 30 mg of DU-176b was administered once daily in the morning in principle for 3 months.
- DU-176b 60 mg: 60 mg of DU-176b was administered once daily in the morning in principle for 3 months.
- Warfarin Potassium: Warfarin was administered once daily at the dose to achieve an INR between 2.0 and 3.0 for 3 months.
Period: Overall Study
Arm/Group | DU176b 30mg | DU-176b 60 mg | Warfarin Potassium
Started | 79 | 80 | 75
Completed | 70 | 68 | 69
Not Completed | 9 | 12 | 6
Not completed — Adverse Event | 2 | 8 | 0
Not completed — Death | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 6 | 3 | 3
Not completed — discontinued before start of treatment | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DU176b 30mg | DU-176b 60 mg | Warfarin Potassium | Total
Number analyzed (Participants) | 79 | 80 | 75 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (9.12) | 65.9 (7.71) | 64.5 (9.51) | 65.1 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 28 | 81
  Male | 51 | 55 | 47 | 153
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 79 | 80 | 75 | 234
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 35 | 35 | 34 | 104
  Singapore | 5 | 4 | 4 | 13
  China | 7 | 8 | 7 | 22
  Korea, Republic of | 32 | 33 | 30 | 95

OUTCOME MEASURES:

1. Primary Outcome: Incidence of All Bleeding
Description: Incidence of all bleeding (major, clinically relevant non-major and minor) in two fixed dosage of DU-176b in comparison with warfarin as active control in subjects with non-valvular AF.
Time Frame: 6 months
Population: The Safety Analysis Set was defined as all subjects who received at least one dose of study drug and had at least one post-dose safety assessment. The primary endpoint were analyzed for the subjects who proceeded to the treatment period in the Safety Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of subjects with bleeds
Arm/Group | DU176b 30mg | DU-176b 60 mg | Warfarin Potassium
Number analyzed (Participants) | 79 | 80 | 75
percentage of subjects with bleeds | 20.3 [12.9 to 30.4] | 23.8 [15.8 to 34.1] | 29.3 [20.2 to 40.4]
Statistical Analysis 1: Comparison: DU176b 30mg vs DU-176b 60 mg; Test type: Superiority or Other; difference in percentages = -3.5, 95% CI 2-sided [-16.2 to 9.4]
Statistical Analysis 2: Comparison: DU176b 30mg vs Warfarin Potassium; Test type: Superiority or Other; difference in percentages = -9.1, 95% CI 2-sided [-22.4 to 4.5]
Statistical Analysis 3: Comparison: DU-176b 60 mg vs Warfarin Potassium; Test type: Superiority or Other; difference in percentage = -5.6, 95% CI 2-sided [-19.3 to 8.2]

2. Secondary Outcome: Evaluation of Incidence of Major Adverse Cardiovascular Events: Stroke, Systemic Embolic Event, Myocardial Infarction, Cardiovascular Death, and Hospitalization for Any Cardiac Condition
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Evaluation of Effects on Biomarkers of Thrombus Formation
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Evaluation of Plasma Concentration of DU-176
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Evaluation of Effects on Pharmacodynamic Biomarkers
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Evaluation of All Clinical and Laboratory Safety Data.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | DU176b 30mg | DU-176b 60 mg | Warfarin Potassium
Serious Adverse Events (participants affected / at risk) | 3/79 | 10/80 | 5/75
Other Adverse Events (participants affected / at risk) | 62/79 | 65/80 | 59/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU176b 30mg (N=79) | DU-176b 60 mg (N=80) | Warfarin Potassium (N=75)
cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Concussion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Back injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU176b 30mg (N=79) | DU-176b 60 mg (N=80) | Warfarin Potassium (N=75)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5)
Gingival bleeding (Gastrointestinal disorders) | 4 (4) | 6 (6) | 0 (0)
Chest discomfort (General disorders) | 4 (4) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 1 (1) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 6 (6) | 5 (5)
Alanine aminotransferase increased (Investigations) | 6 (6) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 9 (9) | 12 (12) | 7 (7)
Diabetes mellitus (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 (6) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7) | 8 (8) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 6 (6) | 2 (2)
Haematuria (Renal and urinary disorders) | 9 (9) | 10 (10) | 14 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 5 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
peptic ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
periodontitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
toothache (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
chest pain (General disorders) | 3 (3) | 1 (1) | 1 (1)
fatigue (General disorders) | 1 (1) | 1 (1) | 2 (2)
influenza (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2)
Blood urea increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Glucose tolerance test abnormal (Investigations) | 1 (1) | 2 (2) | 1 (1)
Hypertriglyceridaemia (Investigations) | 1 (1) | 0 (0) | 2 (2)
myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
flushing (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Korea study sites agree that any results of the study are not to be published individually or collectively in whole or part by study site, its employees or agents until after the coordinated multicenter publication or one year after the termination of the study, whichever occurs fist.